CLINICAL TRIAL: NCT06106308
Title: A Phase 2, Randomized, Open-label Study of Onvansertib in Combination With FOLFIRI and Bevacizumab or FOLFOX and Bevacizumab Versus FOLFIRI and Bevacizumab or FOLFOX and Bevacizumab for First-line Treatment of Metastatic Colorectal Cancer in Patients With a KRAS or NRAS Mutation
Brief Title: Study of Onvansertib in Combination With FOLFIRI and Bevacizumab or FOLFOX and Bevacizumab Versus FOLFIRI and Bevacizumab or FOLFOX and Bevacizumab for First-Line Treatment of Metastatic Colorectal Cancer in Adult Participants With a KRAS or NRAS Mutation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cardiff Oncology (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRDF-004
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colorectal Cancer; CRC; KRAS/NRAS Mutation
Keywords: Metastatic Colorectal Cancer; KRAS Mutation; NRAS Mutation; CRC; First-Line
MeSH Terms: conditions — Colorectal Neoplasms | interventions — onvansertib; IFL protocol; Bevacizumab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Onvansertib 20mg + Standard of Care (Experimental): Participants will receive 20 mg of onvansertib on Days 1 to 5 and Days 15 to 19 of each 28-day treatment cycle + FOLFIRI/BEV on Day 1 and Day 15 of each 28-day treatment cycle.
  Interventions: Drug: Onvansertib; Drug: FOLFIRI; Drug: Bevacizumab
- Onvansertib 30 mg + Standard of Care (SOC) (Experimental): Participants will receive 30 mg of onvansertib + on Days 1 to 5 and Days 15 to 19 of each 28-day treatment cycle + FOLFIRI on Day 1 and Day 15 of each 28-day treatment cycle.
  Interventions: Drug: Onvansertib; Drug: FOLFIRI; Drug: Bevacizumab
- Standard of Care (SOC) (Active Comparator): Participants will receive FOLFIRI/Bev on Day 1 and Day 15 of each 28-day treatment cycle.
  Interventions: Drug: FOLFIRI; Drug: Bevacizumab
- Onvansertib 20 mg + Standard of Care (Experimental): Participants will receive 20 mg of onvansertib on Days 1 to 5 and Days 15 to 19 of each 28-day treatment cycle + FOLFOX on Day 1 and Day 15 of each 28-day treatment cycle.
  Interventions: Drug: Onvansertib; Drug: Bevacizumab; Drug: FOLFOX
- Onvansertib 30 mg + Standard of Care (Experimental): Participants will receive 30 mg onvansertib on Days 1 to 5 and Days 15 to 19 of each 28-day treatment cycle + FOLFOX on Day 1 and Day 15 of each 28-day treatment cycle.
  Interventions: Drug: Onvansertib; Drug: Bevacizumab; Drug: FOLFOX
- Standard of Care (Active Comparator): Participants will receive FOLFOX/Bev on Day 1 and Day 15 of each 28-day treatment cycle.
  Interventions: Drug: Bevacizumab; Drug: FOLFOX

INTERVENTIONS:
Drug: Onvansertib — Oral capsule
  Arms: Onvansertib 20 mg + Standard of Care; Onvansertib 20mg + Standard of Care; Onvansertib 30 mg + Standard of Care; Onvansertib 30 mg + Standard of Care (SOC)
Drug: FOLFIRI — FOLFIRI (irinotecan + fluorouracil [5-FU] + leucovorin) as intravenous (IV) infusion
  Arms: Onvansertib 20mg + Standard of Care; Onvansertib 30 mg + Standard of Care (SOC); Standard of Care (SOC)
Drug: Bevacizumab — IV Infusion
Drug: FOLFOX — FOLFOX (leucovorin + fluorouracil [5-FU] + oxaliplatin) as intravenous (IV) infusion
  Arms: Onvansertib 20 mg + Standard of Care; Onvansertib 30 mg + Standard of Care; Standard of Care

SUMMARY:
The purpose of this study is to assess 2 different doses of onvansertib to select the lowest dose that is maximally effective, and to assess the safety, efficacy, pharmacokinetics, and pharmacodynamics of onvansertib in combination with FOLFIRI + bevacizumab or FOLFOX + bevacizumab in patients with KRAS or NRAS-mutated metastatic colorectal cancer (CRC) in the first-line setting.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic colorectal cancer.
* Documented KRAS or NRAS mutation.
* No previous systemic therapy in the metastatic setting.
* Participants must be willing to submit archival tissue or undergo fresh biopsy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Women of childbearing potential must use contraception or take measures to avoid pregnancy.
* Imaging computed tomography (CT) or magnetic resonance imaging (MRI) of chest/abdomen/pelvis and other scans as necessary to document all sites of disease performed within 28 days prior to the first dose of onvansertib.
* Must have acceptable organ function

Exclusion Criteria:

* Concomitant KRAS or NRAS and BRAF-V600 mutation or microsatellite instability high/deficient mismatch repair.
* Prior treatment with a VEGF inhibitor, including bevacizumab or biosimilars.
* Previous oxaliplatin treatment within 12 months prior to randomization, when arm open.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.
* Anticancer chemotherapy or biologic therapy administered within 28 days prior to the first dose of study drug.
* Untreated or symptomatic brain metastasis.
* Gastrointestinal (GI) disorder(s) that would significantly impede the absorption of an oral agent.
* Unable or unwilling to swallow study drug.
* Uncontrolled intercurrent illness.
* Known hypersensitivity to fluoropyrimidine or leucovorin, irinotecan, or oxalipatin.
* Abnormal glucuronidation of bilirubin; known Gilbert's syndrome.
* Use of strong CYP3A4 or CYP2C19 inhibitors or strong CYP3A4 inducers.
* QTc >470

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 1 year
  ORR defined as the proportion of participants who achieved a best overall Response (BOR) of CR or PR per RECIST Version 1.1 from randomization until disease progression, or death due to any cause, as determined by blinded independent central review.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 1 year
  PFS defined as the time from the date of randomization to the earliest documented disease progression per RECIST version 1.1, or death due to any cause, as determined by blinded independent central review.
Duration of Response (DOR) | Up to approximately 1 year
  DOR defined as the time from the date of first documentation of objective tumor response (CR or PR) to the earliest documented disease progression per RECIST version 1.1, or death due to any cause, as determined by blinded independent central review.
Number of Participants with an Adverse Event (AE) | Up to approximately 1 year
  Type, incidence, causality and severity of AEs based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0. Clinically significant changes from baseline in vital signs, laboratory parameters, electrocardiograms (ECGs), weight, and Eastern Cooperative Oncology Group (ECOG) performance status will be recorded as AEs.
Disease Control Rate (DCR) | Up to approximately 1 year
  DCR defined as CR plus PR plus stable disease (SD), as determined by independent central review.
Overall Survival (OS) | Up to approximately 1 year
  OS defined as the time from drug administration to death due to any cause.
Overall Response (OR) | Up to approximately 1 year
  Defined as CR or PR, PFS, DCR, DOR, and OS associated with a reduction in circulating tumor DNA (ctDNA) mutation allele frequency (MAF).
Maximum Concentration (Cmax) of Onvansertib and metabolites in combination w/FOLFIRI and bevacizumab or FOLFOX and bevacizumab | Day 1 and Day 5 of Cycle 1, and Day 5 of Cycle 3 (cycle is 28 days)
Area Under the Plasma Concentration Curve (AUC) of Onvansertib and metabolites in combination w/FOLFIRI and bevacizumab or FOLFOX and bevacizumab | Day 1 and Day 5 of Cycle 1, and Day 5 of Cycle 3 (cycle is 28 days)
Trough Concentration (Ctrough) of Onvansertib and metabolites in combination w/FOLFIRI and bevacizumab or FOLFOX and bevacizumab | Day 1 and Day 5 of Cycle 1, and Day 5 of Cycle 3 (cycle is 28 days)
Efficacy: Exposure Response Evaluation of Onvansertib | Up to approximately 1 year
Safety: Exposure Response Evaluation of Onvansertib | Up to approximately 1 year

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Pacific Cancer Medical Center, Anaheim, California
  - Comprehensive Blood and Cancer Center - Bakersfield, Bakersfield, California
  - Orange Coast Memorial Medical Center, Fountain Valley, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Department of Medicine-Hematology/Oncology, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - Torrance Memorial Physician Network - Cancer Care and Infusion Center, Torrance, California
  - PIH Health, Whittier, California
  - Memorial Cancer Institute, Hollywood, Florida
  - Mayo Clinic - Florida, Jacksonville, Florida
  - Cleveland Clinic Martin Health, Stuart, Florida
  - Kaiser Permanente, Honolulu, Hawaii
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - The University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Cancer & Hematology Centers of Western Michigan - Lemmen-Holton Cancer Pavilion, Grand Rapids, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Saint Luke's Hospital, Kansas City, Missouri
  - Washington University School of Medicine Center for Advanced Medicine, St Louis, Missouri
  - CCCN, Las Vegas, Nevada
  - Manhattan Hematology Oncology (MHO) Research Foundation, Inc., New York, New York
  - Trihealth Kenwood, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - West Cancer Clinic, Germantown, Tennessee
  - Oncology Consultants, PA, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - VCU Massey Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahn DH, Ridinger M, Cannon TL, Mendelsohn L, Starr JS, Hubbard JM, Kasi A, Barzi A, Samuelsz E, Karki A, Subramanian RA, Yemane D, Kim R, Wu CC, Croucher PJP, Smeal T, Kabbinavar FF, Lenz HJ. Onvansertib in Combination With Chemotherapy and Bevacizumab in Second-Line Treatment of KRAS-Mutant Metastatic Colorectal Cancer: A Single-Arm, Phase II Trial. J Clin Oncol. 2025 Mar;43(7):840-851. doi: 10.1200/JCO-24-01266. Epub 2024 Oct 30. PMID 39475591